CLINICAL TRIAL: NCT03298191
Title: Comparative Study on Tocolysis in Prevention of Preterm Labour
Brief Title: Tocolysis in Prevention of Preterm Labor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed atef mohamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TPL
Record Dates: First submitted 2017-08-26; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Preterm Labor Without Delivery
MeSH Terms: interventions — Magnesium Sulfate; Ritodrine; Calcium Channel Blockers

STUDY DESIGN:
Intervention Model Description: complications ofthe drugs good response to drugs
Who Masked: Participant
Masking Description: false preterm labour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium sulphate (Experimental)
  Interventions: Drug: Magnesium Sulfate
- Ritodrine (Experimental)
  Interventions: Drug: Ritodrine
- Calcium channel blocker (Experimental)
  Interventions: Drug: Calcium Channel Blockers

INTERVENTIONS:
Drug: Magnesium Sulfate — Those women will be given Magnesium Sulfate for tocolysis
  Arms: Magnesium sulphate
Drug: Ritodrine — Those women will be given Ritodrine for tocolysis
  Arms: Ritodrine
Drug: Calcium Channel Blockers — Those women will be given Calcium Channel Blockers for tocolysis
  Arms: Calcium channel blocker

SUMMARY:
Preterm birth is defined as birth before 37 completed weeks of gestation .it occurs in 11.1%of birth globally affecting an estimated 14.9 million babies every year . It is generally accepted that approximately 65%-70%of preterm births are spontaneous,40%-45% of them due to spontaneous preterm labor and 25%-30%following preterm rupture of membranes.preterm birth represents the single largest cause of morbidity and mortality for newborn and is estimated for 29%of deaths in the first four weeks of life and also is estimated for of major cause of morbidity for pregnant women .

Tocolytic agents include a wide range of drugs that can slow or suppress uterine contractions . Tocolytic are considered advantages in spontaneous preterm labor to : (a) allow time for the fetus to mature ,potentially avoiding deleterious effects of pre-maturity . (b)allow time for antenatal corticosteroids to be administered and have clinical effect. (c) allow time for intrauterine transfer to higher-care center where neonatal intensive care facilities are available . the ideal Tocolytic agent should be effective , easy to administer , without significant material ,fetal or neonatal side effects and permit time for antenatal corticosteroids to be administered and take effect . a variety of Tocolytic treatments have been used to inhibit uterine activity in women in spontaneous preterm labor , including betamimetics , calcium channel blockers , magnesium sulfate , prostaglandin inhibitors and oxytocin receptor antagonists however there is considerable global variation in types , doses and regimens of tocolytic agents uses to manage preterm labor .

A comparison study between Ritodrine, magnesium sulfate and Nifedipine in terms of effect and morbidity will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* . Gestational age between 24-37weeks

  * Symptoms such as low backache , cramping ,pelvic pressure, excessive vaginal discharge and vaginal spotting .
  * Regular uterine contractions at least of 30 seconds duration at a rate of more than 4/30 minutes
  * Cervical changes dilatation less than 3cm,effacement lessthan50%.
  * Intact membranes.

Exclusion criteria

* Active vaginal bleeding and placental abruption.
* Chorioamnionitis and intrauterine infection
* Fetal conditions : fetal death or distress, lethal congenital or chromosomal abnormalities and intra uterine growth restriction
* Maternal conditions indicate that pregnancy shouldn't be continued: eclampsia , severe preeclampsia and cardiac diseases
* Drug specific contraindications(contraindication of tocolysis)

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnancy
Enrollment: 300 (Estimated)
Dates: Start 2017-10-25 (Estimated); Primary Completion 2018-04-25 (Estimated); Study Completion 2018-05-25 (Estimated)

PRIMARY OUTCOMES:
The time of delivery | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Atef Mohamed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046